CLINICAL TRIAL: NCT03637972
Title: Clinical Trial to Assess the Removal of Filter Ventilation on Smoking Behavior and Biomarkers
Brief Title: COMET2 Project 1 Filter Ventilation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2018NTLS083; NCT03715491 (obsolete NCT alias)
Record Dates: First submitted 2018-07-12; First posted 2018-08-20 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Smoking; Tobacco Use
Keywords: Cigarette smoking; Filter Ventilation
MeSH Terms: conditions — Smoking; Tobacco Use; Cigarette Smoking | interventions — 3-azido-2,7-naphthalene disulfonate

STUDY DESIGN:
Intervention Model Description: Phase III randomized, open label, multi-center study assessing the impact of filter ventilation. Assigned to ventilated or unventilated cigarettes and either access to ANDS in an experimental marketplace, or no access to ANDS or any other products.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ventilated cigarettes only (Experimental): Filters with approximately 30-36% filter ventilation
  Interventions: Other: Ventilated cigarettes only
- Unventilated cigarettes only (Experimental): Filters with approximately 3.0-4.6% filter ventilation
  Interventions: Other: Unventilated cigarettes only
- Ventilated cigarettes + alternative nicotine delivery systems (Experimental): Filters with approximately 30-36% filter ventilation and access to alternative nicotine delivery systems including e-cigarette/vaping device, medicinal nicotine (lozenge, gum and patch).
  Interventions: Other: Access to Experimental Marketplace: Ventilated cigarettes + alternative nicotine delivery systems
- Unventilated cigarettes + ANDS (Experimental): Filters with approximately 3.0-4.6% filter ventilation and access to alternative nicotine delivery systems including e-cigarette/vaping device, medicinal nicotine (lozenge, gum and patch).
  Interventions: Other: Access to Experimental Marketplace: Unventilated cigarettes + ANDS

INTERVENTIONS:
Other: Ventilated cigarettes only — Participants given vouchers that are exchanged for ventilated cigarettes study cigarettes.
  Arms: Ventilated cigarettes only
Other: Unventilated cigarettes only — Participants given vouchers that are exchanged for unventilated cigarettes study cigarettes.
  Arms: Unventilated cigarettes only
Other: Access to Experimental Marketplace: Ventilated cigarettes + alternative nicotine delivery systems — Participants given vouchers that are exchanged for ventilated cigarettes + alternative nicotine delivery systems cigarettes.
  Arms: Ventilated cigarettes + alternative nicotine delivery systems
Other: Access to Experimental Marketplace: Unventilated cigarettes + ANDS — Participants given vouchers that are exchanged for unventilated cigarettes + ANDS.
  Arms: Unventilated cigarettes + ANDS

SUMMARY:
Phase III randomized, 2 x 2 design, open label, multi-center study that will assess the removal of filter ventilation on smoking behavior and biomarkers in a tobacco and nicotine product marketplace simulation of a real world environment.

DETAILED DESCRIPTION:
This randomized, open label, controlled multi-site study will simulate a "real world" tobacco environment by providing access to an experimental marketplace where they will be given vouchers that can be exchanged for assigned study cigarettes (either ventilated or unventilated) and two of the groups will also have access to non-combusted tobacco/nicotine products.

Subjects (N=550; N=125 in each group) will be randomly assigned to: 1) Ventilated cigarettes only; or 2) Unventilated cigarettes only; 3) Ventilated cigarettes + alternative nicotine delivery systems (ANDS); 4) Unventilated cigarettes + ANDS.

Smokers will undergo an in person screening and then a 12 week experimental trial consisting of 2 weeks of baseline; 2 weeks of usual brand cigarettes in the marketplace and 8 weeks on the study cigarettes in the marketplace, plus a follow-up visit 4 weeks after the intervention is over. The experimental period will simulate a "real world" environment by providing participants with vouchers for a specified number of points that can be exchanged for study cigarettes and/or ANDS. At the end of the study they can exchange unspent points for money.

Biomarker samples (total nicotine equivalents, tobacco specific nitrosamines, volatile organic compound and inflammation markers), smoking topography and inhalation measures are taken at baseline and end of trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Biochemically confirmed regular cigarette smoker

Exclusion Criteria:

* Unstable health
* Unstable medications
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
The total NNAL at Week 8 Visit | Week 8
  The total NNAL at the 8 week visit of Phase 3 adjusted for NNAL at baseline (Phase 2, week 00)
Mean CPD based on 7 day IVR before week 8 visit. | Week 8
  The mean CPD based on 7 days IVR data before week 8 visit adjusted for the mean CPD during Phase 2, week 00.

SECONDARY OUTCOMES:
Change in biomarkers (TNE, NNN, mercapturic acids, PheT) from baseline | Week 8
  Absolute change from baseline in other biomarkers (e.g., TNE, NNN, mercapturic acids, PheT)
Number of cigarette-free days | Week 8
  number of cigarette-free days based on no cigarettes smoked in the previous day on IVR (dropouts with no IVR data are assumed to be smoking)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Hatsukami, Ph.D, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Tobacco Research Program, Minneapolis, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Intend to share findings from this research through publications and presentations. Institutions and individuals wishing to access any resources or data must contact the Principal Investigator (Hatsukami). Data generated by this grant will be made to outside investigators, according to NIH Guidance. When data are shared, there will be no limits placed on how the data will be used. Users will agree, however, that the recipient must not transfer the data to other users and that the data are only to be used for research purposes. A record of transfer of data and a copy of the dataset that was distributed will be kept by University of Minnesota.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will not be available until primary and secondary papers are accepted for publication.
Access Criteria: Persons requesting data must do so in writing, identifying their affiliation and how the data will be used. Upon review, access will be determined.